CLINICAL TRIAL: NCT00946387
Title: A Relative Bioavailability Study of Ondansetron HCl 24 mg Tablets Under Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability Study of Ondansetron HCl 24 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B043712
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Nausea; Vomiting
Keywords: Antiemetic
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron; halofantrine

ARMS (2):
- 1 (Experimental): Ondansetron HCl 24 mg Tablets (Sandoz, Inc.)
  Interventions: Drug: Ondansetron HCl 24 mg Tablets (Sandoz, Inc.)
- 2 (Active Comparator): Zofran (Ondansetron HCl) 24 mg Tablets (GlaxoSmithKline)
  Interventions: Drug: Zofran (Ondansetron HCl) 24 mg Tablets (GlaxoSmithKline)

INTERVENTIONS:
Drug: Ondansetron HCl 24 mg Tablets (Sandoz, Inc.)
  Arms: 1
Drug: Zofran (Ondansetron HCl) 24 mg Tablets (GlaxoSmithKline)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability study of Ondansetron HCl 24 mg tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 22 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-09; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong, M.D., Principal Investigator — Novum Pharmaceutical Research Services